

#### Protocol C4891008

An Interventional, Phase 1, Open-Label, Fixed-Sequence, 2-Period Study to Evaluate the Effect of a Single Oral Dose of ARV-471 (PF-07850327) on the Pharmacokinetics of Dabigatran in Healthy Participants

Statistical Analysis Plan (SAP)

Version: 1

**Date:** 17 Jan 2023

# TABLE OF CONTENTS

| LIST OF TABLES | 4 |
|-------------------------------------------------------------------|----|
| APPENDICES | 4 |
| 1. VERSION HISTORY | 5 |
| 2. INTRODUCTION | 5 |
| 2.1. Modifications to the Analysis Plan Described in the Protocol | 5 |
| 2.2. Study Objectives, Endpoints, and Estimands | 5 |
| 2.3. Study Design | 6 |
| 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 7 |
| 3.1. Primary Endpoints | 7 |
| 3.2. Secondary Endpoints | 9 |
| 3.3. Other Endpoints | 9 |
| 3.4. Baseline Variables | 9 |
| 3.5. Safety Endpoints | 9 |
| 3.5.1. Adverse Events | 9 |
| 3.5.2. Laboratory Data | 9 |
| 3.5.3. Vital Signs. | 10 |
| 3.5.4. Electrocardiograms. | 10 |
| 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS) | 10 |
| 5. GENERAL METHODOLOGY AND CONVENTIONS | 11 |
| 5.1. Hypotheses and Decision Rules. | 11 |
| 5.2. General Methods | 11 |
| 5.2.1. Analyses for Binary/Categorical Endpoints | 11 |
| 5.2.2. Analyses for Continuous Endpoints | 11 |
| 5.3. Methods to Manage Missing Data | 11 |
| 5.3.1. Pharmacokinetic Data | 11 |
| 5.3.2. Safety Data | 12 |
| 6. ANALYSES AND SUMMARIES | 13 |
| 6.1. Primary Endpoints | 13 |
| 6.2. Secondary Endpoints | 13 |
| 6.3. Other Endpoints | 13 |

| 6.4. Subset Analyses | 15 |
|-------------------------------------------------------|----|
| 6.5. Baseline and Other Summaries and Analyses | 15 |
| 6.5.1. Demographic Summaries | 15 |
| 6.5.2. Study Conduct and Participant Disposition | 15 |
| 6.5.3. Study Treatment Exposure | 15 |
| 6.5.4. Concomitant Medications and Nondrug Treatments | 15 |
| 6.6. Safety Summaries and Analyses | 15 |
| 6.6.1. Adverse Events | 15 |
| 6.6.2. Laboratory Data | 16 |
| 6.6.3. Vital Signs | 16 |
| 6.6.4. Electrocardiograms | 16 |
| 7. INTERIM ANALYSES | 16 |
| 7.1. Introduction | 16 |
| 7.2. Interim Analyses and Summaries | 16 |
| ADDENDICES | 17 |

## LIST OF TABLES

| Table 1. Summary of Changes | 5 |
|-------------------------------------------------------|-----|
| Table 2. Plasma PK Parameters | 8 |
| Table 3. PK Parameters to be Summarized Descriptively | 14 |
| APPENDICES | |
| | 1.7 |
| Appendix 1. SAS Code for Analyses | 17 |
| Appendix 2. List of Abbreviations | 18 |

NOTE: Italicized text within this document has been taken verbatim from the Protocol.

#### 1. VERSION HISTORY

**Table 1. Summary of Changes** 

| Version/<br>Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1 /<br>17 Jan 2023 | Original<br>04 Nov 2022 | N/A | N/A |

#### 2. INTRODUCTION

ARV-471 (PF-07850327) is a potent, selective, orally bioavailable PROTAC® small molecule that induces degradation of the ER. ARV-471 is a hetero-bifunctional PROTAC molecule that simultaneously binds the ER and the cereblon E3 ligase complex, enabling protein-protein interactions between ER and the ligase complex. As a result, the ER becomes polyubiquitinated on accessible lysine residues and subsequently undergoes targeted degradation by the proteasome.

Based on available data, it is possible that administration of a P-gp substrate, dabigatran etexilate (as mesylate), with ARV-471 may lead to increased plasma exposures of dabigatran (active drug). The purpose of this study is to estimate the effect of ARV-471 on the PK of dabigatran in healthy participants.

This SAP provides the detailed methodology for summary and statistical analyses of the data collected in Study C4891008.

## 2.1. Modifications to the Analysis Plan Described in the Protocol

None.

## 2.2. Study Objectives, Endpoints, and Estimands

The following are the objectives and endpoints in this study. Estimand framework will not be applied to this Phase 1 study in healthy participants.

| Objectives | Endpoints |
|---|---|
| Primary: | Primary: |
| • To estimate the effect of a single oral 200 mg dose of ARV-471 on the single dose pharmacokinetic of dabigatran in healthy participants. | • Plasma total dabigatran (sum of unconjugated and glucuronide-conjugated dabigatran) PK parameters alone and following administration of a single 200 mg dose of ARV-471: C <sub>max</sub> , AUC <sub>inf</sub> (AUC <sub>last</sub> if AUC <sub>inf</sub> cannot be estimated). |
| Secondary: | Secondary: |
| • To evaluate the safety and tolerability of dabigatran etexilate (as mesylate) alone and following administration with a single 200 mg dose of ARV-471 | Safety: TEAEs, clinical laboratory tests,<br>vital signs, PE, and ECGs |
| Other: | Other: |
| · CCI | |

### 2.3. Study Design

This will be a Phase 1, open-label, 2-period, fixed sequence study to estimate the effect of a single oral ARV-471 dose on the PK of a P-gp substrate, dabigatran etexilate (as mesylate), in healthy male participants or healthy female participants of nonchildbearing potential. An attempt will be made to enroll more than 50% participants as female participants with nonchildbearing potential in this study since ARV-471 is being developed for the treatment in a population that is predominately female.

This study will consist of 2 periods with a fixed sequence treatment design. On Period 1 Day 1, a standard breakfast will be provided prior to dosing. The standard breakfast will be completely consumed within an approximately 20-minute period. A single dose of 75 mg dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) will be administered approximately 2 hours (120 minutes) after starting the standard breakfast. To adequately remove any drug effects of dabigatran, a minimum washout period of 4 days is followed after dabigatran etexilate (as mesylate) administration on Period 1 Day 1.

On Period 2 Day 1, a standard breakfast will be provided prior to ARV-471 and dabigatran etexilate (as mesylate) dosing. The standard breakfast will be completely consumed within an

approximately 20-minute period. A single dose of 200 mg ARV-471 (as 2 tablets of 100 mg) will be administered approximately 10 minutes after the completion of the breakfast. A single dose of 75 mg dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) will be administered approximately 1.5 hour (90 minutes) after the start of ARV 471 dosing, which is approximately 2 hours (120 minutes) after the start of the breakfast.

A sufficient number of participants will be screened to ensure that at least 24 participants will be enrolled in the study. Participants who withdraw may be replaced at the discretion of the sponsor. Healthy participants will be screened to determine eligibility within 28 days prior to study treatment (ie, within 28 days prior to Day 1 of Period 1). Medical history and results of physical examination, physical measurements, vital signs, 12-lead ECGs, and clinical laboratory evaluations will determine eligibility.

Participants will report to the CRU at least 12 hours prior to Day 1 dosing in Period 1 and will be required to stay in the CRU for 8 days and 7 nights. Washout period will begin after the first dose of study treatment.

| Fixed-<br>Sequence | Period 1 | | Period 2 | |
|---|---|---|---|---|
| Screening | Day 1-4 | At least 4-Day<br>washout | Day 1- 3 | Follow-up |
| All screening<br>should be done<br>2 to 28 days<br>before the first<br>dose | (Reference) 75 mg single oral dose of dabigatran etexilate (as mesylate) administered approximately 2 hours (120 minutes) after the start of a standard breakfast (Period 1 Day 1) | The washout will<br>begin after the<br>first dose of<br>study medication | (Test) 200 mg single oral dose of ARV-471 administered approximately 30 minutes after the start of the standard breakfast and 75 mg single oral dose of dabigatran etexilate (as mesylate) administered approximately 1.5 hours (90 minutes) after the start of ARV-471 dosing, which is approximately 2 hours (120 minutes) after the start of the breakfast (Period 2 Day 1). | Follow-up must<br>occur 28 to<br>35 days after<br>administration<br>of the final<br>dose of study<br>intervention |

# 3. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

#### 3.1. Primary Endpoints

The primary endpoints of the study are plasma AUC<sub>inf</sub> (if data permit, otherwise AUC<sub>last</sub>) and C<sub>max</sub> of total dabigatran (sum of uncongugated and glucuronide-congugated dabigatran) alone and following administration of a single 200 mg dose of ARV-471. Adjusted geometric mean ratios of AUC<sub>inf</sub> (if data permit, otherwise AUC<sub>last</sub>) and C<sub>max</sub> will be derived.

The plasma PK parameters for total dabigatran will be derived (as data permit and as appropriate) from the concentration time profiles as detailed in Table 2 for each analyte and treatment. Actual PK sampling times will be used in derivation of PK parameters. In the case that actual PK sampling times are not available, nominal PK sampling time will be used in the derivation of PK parameters.

Table 2. Plasma PK Parameters

| Parameter <sup>a</sup> | Analyte | Definition | Method of Determination |
|---|---|---|---|
| AUClast | total dabigatran, | Area under the plasma concentrationtime profile from time 0 to the time of last quantifiable | Linear/Log trapezoidal method. |
| AUC a inf | total dabigatran, | concentration (C <sub>last</sub> ).<br>Area under the plasma | $AUC_{last} + (C_{last}^*/k_{el}),$ |
| | CCI | concentrationtime<br>profile from time 0<br>extrapolated to infinite<br>time. | where $C_{last}^*$ is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis. |
| $C_{max}$ | total dabigatran, | Maximum plasma concentration | Observed directly from the data. |
| C <sub>last</sub> | total dabigatran, | Last measurable observed concentration | Observed directly from the data. |
| T <sub>max</sub> | total dabigatran, | Time for C <sub>max</sub> | Observed directly from the data. |
| T <sub>last</sub> | total dabigatran, | Time for C <sub>last</sub> | Observed directly from the data. |
| $t_{\frac{a}{\frac{1}{2}}}$ | total daoigatran, | Terminal elimination | $Log_{e}(2)/k_{el}$ , where $k_{el}$ is the terminal phase |
| | CCI | half-life | rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline will be used in the regression. |
| CL/F <sup>a</sup> | total dabigatran, | Apparent clearance | Dose/(AUCinf) |
| CCI | | | |
| CCI | | | |
| | | | AAx — |
| | | | AAX |

a. if data permits and as appropriate.

## 3.2. Secondary Endpoints

The secondary endpoints are the overall safety profile of dabigatran etexilate (as mesylate) alone and following administration with a single 200 mg dose of ARV-471, as characterized by adverse events, laboratory tests, vital signs, and ECGs (discussed in Section 3.5).

## 3.3. Other Endpoints



In addition, other total dabigatran PK parameters ( $C_{last}$ ,  $AUC_{last}$ ,  $T_{max}$ ,  $T_{last}$ ,  $t_{1/2}$ , CL/F,  $V_z/F$ , as data permit) will also be derived following the methodology described above.

#### 3.4. Baseline Variables

Baseline participant characteristics will be collected according to the schedule of activities (SoA) as specified in the protocol.

## 3.5. Safety Endpoints

The following data will be considered in standard safety summaries (see protocol for collection days, baseline assessment, and list of parameters):

- Adverse events (AE)
- Laboratory data
- Vital signs data
- ECG results

## 3.5.1. Adverse Events

Any adverse event occurring following start of treatment will be considered a treatment emergent adverse event (TEAE). Events that occur during follow-up within the lag time of up to 28 days after the last dose of study intervention will be counted as treatment emergent and attributed to the last treatment taken. Events that occur during the washout period between study periods will be counted as treatment emergent and attributed to the previous treatment taken. The time period for collecting AEs ("active collection period") for each participant begins from the time the participant provides informed consent.

#### 3.5.2. Laboratory Data

Safety laboratory tests will be performed as described in the protocol. To determine if there are any clinically significant laboratory abnormalities, the haematological, clinical chemistry

(serum) and urinalysis safety tests will be assessed against the criteria specified in the sponsor reporting standards. The assessment will not take into account whether each participant's baseline test result is within or outside the laboratory reference range for the particular laboratory parameter.

For both Periods, the baseline measurement is the predose measurement on Period 1 Day -1. Changes from baseline will be defined as the change between the baseline and postdose measurements.

## 3.5.3. Vital Signs

Supine blood pressure (BP) and pulse rate (PR) will be measured at times specified in the SoA in the protocol.

For both Periods, the baseline measurement is the predose measurement on Period 1 Day 1. Changes from baseline will be defined as the change between the baseline and postdose measurements.

## 3.5.4. Electrocardiograms

QT interval, QTcF, PR, QRS and heart rate (HR) will be recorded at each assessment time indicated in the SoA given in the protocol. If not supplied, QTcF will be derived using Fridericia's heart rate correction formula:

$$QTcF = QT / (RR)^{(1/3)}$$
 where  $RR = 60/HR$  (if not provided)

For both Periods, the baseline value is the average of the triplicate ECG measurements collected before dose administration on Period 1 Day 1. Changes from baseline will be defined as the change between the baseline ECG and the postdose ECG measurement.

The maximum absolute value (postdose) and the maximum increase from baseline for QTcF over all measurements taken postdose will be determined.

The maximum increase from baseline will be calculated by first subtracting the baseline value from each postdose measurement to give the change from baseline. The maximum of these values over the respective period will then be selected, except in the case where a participant does not show an increase. In such an instance, the minimum decrease should be taken.

#### 4. ANALYSIS SETS (POPULATIONS FOR ANALYSIS)

Data for all participants will be assessed to determine if participants meet the criteria for inclusion in each analysis population prior to releasing the database. Classifications will be documented per standard operating procedures.

| Participant Analysis Set | Description |
|---|---|
| Enrolled | "Enrolled" means a participant's, or their legally authorized representative's, agreement to participate in a clinical study following completion of the informed consent process and assigned to study intervention. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. |
| Safety Analysis Set | All participants who have received at least 1 dose of study intervention. Participants will be analyzed according to the product they actually received. |
| PK Concentration Set | All participants who are in the Safety Analysis Set and have at least 1 measurable concentration of CCI. |
| PK Parameter Set | All participants who are in the Safety Analysis Set and have at least 1 PK parameter of interest for CCI. |

#### 5. GENERAL METHODOLOGY AND CONVENTIONS

Final analysis will be performed after study participant data set release following last participant last visit.

## 5.1. Hypotheses and Decision Rules

No statistical hypothesis will be tested in this study.

#### 5.2. General Methods

## 5.2.1. Analyses for Binary/Categorical Endpoints

For binary or categorical variables, number of participants, numbers and percentages of participants meeting the categorical criteria will be presented in accordance with the Clinical Data Interchange Standards Consortium and Pfizer Standards (CaPS).

#### **5.2.2.** Analyses for Continuous Endpoints

For continuous variables, the data will be summarized using the number of participants, mean, median, standard deviation (SD), minimum, and maximum in accordance with the CaPS. For appropriate PK parameters, geometric mean and geometric coefficient of variation (%CV) will also be summarized.

## 5.3. Methods to Manage Missing Data

#### 5.3.1. Pharmacokinetic Data

Methods to handle missing PK data are described below.

## **Concentrations Below the Limit of Quantification:**

In all data presentations except listings, concentrations below the limit of quantification (BLQ) will be set to zero. In listings BLQ values will be reported as "<LLQ", where LLQ will be replaced with the value for the lower limit of quantification.

## **Deviations, Missing Concentrations and Anomalous Values:**

In summary tables and plots of median profiles, statistics will be calculated having set concentrations to missing if one of the following cases is true:

- 1. A concentration has been collected as ND (ie, not done) or NS (ie, no sample).
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged as anomalous by the pharmacokineticist.

Summary statistics will not be presented at a particular time point if more than 50% of the data are missing.

An anomalous concentration value is one that, after verification of bioanalytical validity, is grossly inconsistent with other concentration data from the same individual or from other participants. For example, a BLQ concentration that is between quantifiable values from the same dose is considered as anomalous. Anomalous concentration values may be excluded from PK analysis at the discretion of the PK analyst or pharmacokineticist.

#### **PK Parameters:**

Actual PK sampling times will be used in the derivation of PK parameters. If a PK parameter cannot be derived from a participant's concentration data, the parameter will be coded as NC (not calculated; NC values will not be generated beyond the day that a participant discontinues). In summary tables, statistics will be calculated by setting NC values to missing; and statistics will be presented for a particular treatment with ≥3 evaluable measurements. PK parameter analyses will not be performed for a particular parameter if more than 50% of the data are NC.

If an individual participant has a known biased estimate of a PK parameter (due for example to an unexpected event such as vomiting before all the compound is adequately absorbed from the gastrointestinal tract), this will be footnoted in summary tables and will not be included in the calculation of summary statistics or statistical analyses.

## 5.3.2. Safety Data

Missing values in standard summaries of AEs, laboratory data, vital signs, and ECGs will be imputed according to CaPS.

#### 6. ANALYSES AND SUMMARIES

## 6.1. Primary Endpoints

The primary endpoints plasma AUC<sub>inf</sub> (if data permit, otherwise AUC<sub>last</sub>) and C<sub>max</sub> of total dabigatran (sum of uncongugated and glucuronide-congugated dabigatran) alone and following administration of a single 200 mg dose of ARV-471 will be summarized descriptively by treatment and will include the set of summary statistics as specified in Table 3.

Total dabigatran PK parameters following a single dose administration will be derived from the plasma concentration versus time profiles using non-compartmental methods, as data permit and as appropriate. The plasma concentrations of total dabigatran will be listed and descriptively summarized by nominal PK sampling time and treatment. Individual participant, as well as mean and median profiles of the plasma concentration time data will be plotted by treatment for each analyte using actual (for individual) and nominal (for mean and median) times respectively. Mean and median profiles will be presented on both linear and semi-log scales. For comparison of total dabigatran only, AUC<sub>inf</sub> (as data permit), AUC<sub>last</sub>, and C<sub>max</sub> with and without ARV-471, box and whisker plots of these parameters will be plotted by treatment for each analyte.

Natural log transformed parameters (AUC<sub>inf</sub> [if data permit], AUC<sub>last</sub>, and C<sub>max</sub>) of total dabigatran (sum of unconjugated or glucuronide-conjugated dabigatran) will be analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs will be obtained from the model. The adjusted mean differences and 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CI for the ratios. Dabigatran administered alone will be the reference treatment and ARV-471 co-administered with dabigatran will be the test treatment.

Residuals from the model will be examined for normality and the presence of outliers via visual inspection of plots of residuals vs predicted values and normal probability plots of residuals but these will not be included in the CSR. If there are major deviations from normality or outliers then the effect of these on the conclusions will be investigated through alternative transformations and/or analyses excluding outliers. Justification for any alternative to the planned analysis will be provided in the clinical study report.

## 6.2. Secondary Endpoints

Safety data will be analyzed in accordance with the CaPS (see Section 6.6).



Table 3. PK Parameters to be Summarized Descriptively

| Parameter | Summary Statistics |
|---|---|
| AUCinf, AUClast, Cmax, | N, arithmetic mean, median, SD, %CV, minimum, maximum, geometric mean and geometric %CV |
| T <sub>max</sub> , T <sub>last</sub> | N, median, minimum, maximum |
| t <sub>1/2</sub> | N, arithmetic mean, median, SD, %CV, minimum, maximum |

For comparison of total dabigatran only, AUC<sub>inf</sub> (as data permit), AUC<sub>last</sub>, and C<sub>max</sub> with and without ARV-471, box and whisker plots will be plotted as detailed in Section 6.1 under primary endpoints.

Supporting data from the estimation of t<sub>1/2</sub> and AUC<sub>inf</sub> will be listed by analyte and treatment: terminal phase rate constant (k<sub>el</sub>); goodness of fit statistic from the log-linear regression (r<sup>2</sup>); the percent of AUC<sub>inf</sub> based on extrapolation (AUC<sub>extrap%</sub>); and the first, last, and number of time points used in the estimation of K<sub>el</sub>. These data may be included in the clinical study report.

#### PK concentration summaries:

The plasma concentrations of Colombia will be listed and descriptively summarized by nominal PK sampling time and treatment (dabigatran etexilate alone in Period 1, and dabigatran etexilate following administration of ARV-471 in Period 2) for the PK Concentration Analysis Set. Individual participant and summary profiles (mean and median plots) of the plasma concentration-time data will be plotted by treatment using actual and nominal times, respectively. Mean and median plasma concentration profiles will be presented on both linear and semi-log scales.

Presentations for plasma concentrations for each analyte will include:

- A listing of all concentrations sorted by participant ID, period, treatment and nominal time postdose. The concentration listing will also include the actual times. Deviations from the nominal time will be provided in a separate listing.
- A summary of concentrations by treatment and nominal time postdose, where the set of statistics will include n, mean, median, SD, %CV, minimum, maximum and the number of concentrations above the LLQ.
- Median concentrations time plots (on both linear and semi-log scales) against nominal time postdose by treatment (all treatments on the same plot per scale, based on the summary of concentrations by treatment and time postdose).

- Mean concentrations time plots (on both linear and semi-log scales) against nominal time
  postdose by treatment (all treatments on the same plot per scale, based on the summary of
  concentrations by treatment and time postdose).
- Individual concentration time plots by treatment (on both linear and semi-log scales) against actual time postdose (there will be separate spaghetti plots for each treatment per scale).
- Individual concentration time plots by participant (on both linear and semi-log scales) against actual time postdose [there will be separate plots for each participant (containing all treatments) per scale].

## 6.4. Subset Analyses

There are no planned subset analyses.

## 6.5. Baseline and Other Summaries and Analyses

## 6.5.1. Demographic Summaries

Demographic characteristics will be summarized for enrolled population in accordance with the CaPS.

## 6.5.2. Study Conduct and Participant Disposition

Participants evaluation groups will show end of study participant disposition. Frequency counts will be supplied for participant discontinuation(s) by treatment (dabigatran etexilate alone in Period 1, and dabigatran etexilate following administration of ARV-471 in Period 2). Data will be reported in accordance with the CaPS.

## 6.5.3. Study Treatment Exposure

Study treatment exposure will be listed.

#### 6.5.4. Concomitant Medications and Nondrug Treatments

All concomitant medication(s) as well as non-drug treatment(s) will be reported in the listings.

### 6.6. Safety Summaries and Analyses

All safety analyses will be performed on the Safety Analysis Set.

Safety data will be presented in tabular and/or graphical format and summarized descriptively, where appropriate.

#### 6.6.1. Adverse Events

Adverse events will be reported in accordance with the CaPS.

Participant discontinuations due to adverse events will be detailed by treatment. Data will be reported in accordance with the CaPS.

## 6.6.2. Laboratory Data

Laboratory data will be listed and summarized by treatment in accordance with the CaPS.

## 6.6.3. Vital Signs

Vital signs data will be listed and summarized by treatment in accordance with the CaPS.

## 6.6.4. Electrocardiograms

Changes from baseline for the ECG parameters HR, QTcF, PR interval, and QRS complex will be summarized by treatment and time. The frequency of uncorrected QT values above 500 ms will be tabulated.

The number (%) of participants with maximum postdose QTcF values and maximum increases from baseline in the following categories will be tabulated by treatment:

## Safety QTcF Assessment

| Degree of | Mild (ms) | Moderate (ms) | Severe (ms) |
|------------------------|-----------|---------------|-------------|
| Prolongation | | | |
| Absolute value | >450-480 | >480-500 | >500 |
| Increase from baseline | | 30-60 | >60 |

#### 7. INTERIM ANALYSES

No formal interim analysis will be conducted for this study. As this is an open-label study, the sponsor may conduct unblinded reviews of the data during the course of the study for the purpose of safety assessment, facilitating PK modeling, and/or supporting clinical development.

#### 7.1. Introduction

Not applicable.

## 7.2. Interim Analyses and Summaries

Available safety and PK data may be reviewed.

## **APPENDICES**

## **Appendix 1. SAS Code for Analyses**

An example of the PROC MIXED code is provided below:

## For the primary objective:

• Treatment B (Test) vs Treatment A (Reference)

```
proc mixed data=tab.pk;
    class trt participant;
    model l&var=trt / ddfm=KR;
    random participant / subject=participant;
    lsmeans trt;
    estimate 'B vs A' trt -1 1 /cl alpha=0.1;

    ods 'Estimates' out=est&var;
    ods 'Ismeans' out=ls&var;
    ods 'covparms' out=cov&var;
    ods 'tests3' out=tst&var;
run;

/* Letter assignments for treatments (trt) within the estimate statement above are as follows
A: single dose of dabigatran etexilate 75 mg
B: single dose of 200 mg ARV-471 + single dose of dabigatran etexilate 75 mg
*/
```

# Appendix 2. List of Abbreviations

| Abbreviation | Term |
|---|---|
| %CV | coefficient of variation |
| AE | adverse event |
| ANOVA | analysis of variance |
| AUCextrap% | the percent of AUC <sub>inf</sub> based on extrapolation |
| AUCinf | area under the plasma concentration-time profile from time zero |
| | extrapolated to infinite time |
| AUClast | area under the plasma concentration-time profile from time zero to |
| | the time of the last quantifiable concentration |
| BLQ | below the limit of quantitation |
| BP | blood pressure |
| CaPS | Clinical Data Interchange Standards Consortium and Pfizer |
| | Standards |
| CI | confidence interval |
| CL/F | apparent clearance |
| Clast | last measurable observed concentration |
| Cmax | maximum plasma concentration |
| CRF | case report form |
| CSR | clinical study report |
| CYP3A | cytochrome P450, family 3, subfamily A |
| ECG | electrocardiogram |
| ER | estrogen receptor |
| HR | heart rate |
| kel | elimination rate constant estimated from the log-linear regression |
| | analysis |
| LLQ | lower limit of quantitation |
| ms | milliseconds |
| CCI | |
| N/A | not applicable |
| NC | not calculated |
| ND | not done |
| NS | no sample |
| P-gp | p-glycoprotein |
| PK | pharmacokinetic(s) |
| PR | pulse rate |
| QRS | Combination of Q-, R- and S- wave on an electrocardiogram |
| | representing ventricular depolarization |
| QTc | corrected QT |
| QTcF | corrected QT (Fridericia method) |

| Abbreviation | Term |
|-------------------|----------------------------------------------------------|
| $\mathbf{r}^2$ | goodness of fit statistic from the log-linear regression |
| rBA | relative bioavailability |
| RR | respiratory rate |
| SAP | statistical analysis plan |
| SD | standard deviation |
| SoA | schedule of activities |
| t <sub>1/2</sub> | terminal plasma elimination half-life |
| TEAE | treatment emergent adverse event |
| Tlast | time for C <sub>last</sub> |
| Tmax | time for C <sub>max</sub> |
| V <sub>z</sub> /F | apparent volume of distribution after oral dose |